CLINICAL TRIAL: NCT01670890
Title: Efficacy and Safety of Salvage Treatment With Dose-dense TMZ Plus CDDP in the Patients With Recurrent Malignant Gliomas: a Multicentre,Prospective Clinical Study
Brief Title: Efficacy and Safety of TMZ Plus CDDP in the Patients With Recurrent Malignant Gliomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Tianjin Medical University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pumch-neurosurgery-01
Record Dates: First submitted 2012-08-19; First posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Malignant Gliomas
Keywords: temozolomide(TMZ); cisplatin(CDDP); recurrent malignant gliomas
MeSH Terms: conditions — Glioma | interventions — Temozolomide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TMZ group (Active Comparator): patients were treated with TMZ alone
  Interventions: Drug: TMZ
- TMZ plus CDDP group (Experimental): patients were treated with TMZ plus CDDP
  Interventions: Drug: TMZ plus CDDP

INTERVENTIONS:
Drug: TMZ — patients were treated with TMZ alone,Oral TMZ 50mg/m2/day,day 1 to 28,for 6 cycles
  Other Names: temozolomide
  Arms: TMZ group
Drug: TMZ plus CDDP — patients were treated with TMZ plus CDDP,CDDP was administered iv from day 1 to 3 with the total dose of 100mg and TMZ was administered orally 50mg/m2/day,day 1 to 28,for 6 cycles
  Other Names: temozolomide and cisplatin
  Arms: TMZ plus CDDP group

SUMMARY:
Temozolomide is the standard adjuvant chemotherapy of newly-diagnosis malignant gliomas.Cisplatin , a kind of chemotherapeutics, can enforce the anti-tumor effects of TMZ. Up to now, the prognosis of recurrent gliomas is very pessimistic and the standard treatment procedure has not been established yet.

The prospective,multicentre phase II clinical study is to evaluate the efficacy and safety of TMZ and CDDP in patients with recurrent malignant gliomas

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age>=18 and <=70years old
* Histological diagnosis of malignant gliomas(WHO III or IV)
* The status of methylation of promotor of MGMT should be detected.
* The time to be enrolled should be more than 90 days after the irradiation.
* The patients with recurrent gliomas were treated with non-dose-dense TMZ therapy before enrollment.
* Performance status(Karnofsky index)>=60
* Life expectancy more than 3 months

Exclusion Criteria:

* Ages:< 18 years or > 70 years
* Abnormal function of liver or renal(value more than 1.5 fold normal upper limit )
* Blood routing: Hb < 100g/l， WBC < 4.0×109/l; PLT < 100×109/l
* Pregnant or lactating women
* Allergic to administered drugs
* Radiation treatment in the previous 90 days or stereotactic radiation surgery within 60 days before enrollment
* The patients with recurrent gliomas were treated with dose-dense TMZ therapy before enrollment.
* Life expectancy less than 3 months
* Participation in other clinical trials in the 90previous days before enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
over all survival | 1 year

SECONDARY OUTCOMES:
progression free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: wang renzhi, MD, Study Chair — Peking Union Medical College Hospital
Locations (3):
- China (3):
  - Beijing Tiantan Hospital Affiliated to Capital Medial University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Tianjin medical university general university, Tianjin, Tianjin Municipality